CLINICAL TRIAL: NCT02262169
Title: DLBS2411 Treatment for Ulcer Healing in Non-Bleeding Peptic Ulcers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated due to internal technical issues at study site
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS2411-0313
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Non-Bleeding Peptic Ulcers
Keywords: Non-Bleeding Peptic Ulcers, DLBS2411, Ulcer Healing
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment I (Active Comparator): 2 Omeprazole capsules 20 mg once daily and 1 placebo caplet of DLBS2411, twice daily
  Interventions: Drug: Omeprazole; Drug: Placebo caplet of DLBS2411
- Treatment II (Experimental): 1 DLBS2411 caplet 250 mg twice daily and 2 placebo capsules of Omeprazole once daily
  Interventions: Drug: DLBS2411; Drug: Placebo capsule of Omeprazole

INTERVENTIONS:
Drug: Omeprazole — 2 Omeprazole capsules 20 mg, once daily
  Arms: Treatment I
Drug: Placebo caplet of DLBS2411 — 1 placebo caplet of DLBS2411, twice daily
  Other Names: Placebo caplet of Redacid
  Arms: Treatment I
Drug: DLBS2411 — 1 DLBS2411 caplet 250 mg, twice daily
  Other Names: Redacid
  Arms: Treatment II
Drug: Placebo capsule of Omeprazole — 2 placebo capsules of Omeprazole, once daily
  Arms: Treatment II

SUMMARY:
This is a 2-arm, prospective, double-blind, double-dummy, randomized-controlled study using DLBS2411 at a dose of 250 mg twice daily (before morning and evening meals), or omeprazole at a dose of 40 mg once daily (before morning meal), for an 8-week course of therapy, for the treatment of patients with any non-bleeding peptic ulcers.

DLBS2411 is a bioactive fraction of an Indonesian native herbal, Cinnamomum burmanii, locally known as kayu manis have been proven at cellular and genetic levels to have an antiulcer effect through both suppressing the gastric acidity and enhancing gastric mucosal protection. The anti-secretory effect of DLBS2411 is exerted through the inhibition of H+/K+ ATPase 'pump' as well as down-regulation of the H+/K+ ATPase gene expression, thus suppressing gastric acid secretion; while its gastro-protective defense mechanism works through the promotion of COX-2 derived prostaglandin (PgE2) synthesis, stimulating gastric-epithelial mucous and bicarbonate secretion; anti-oxidative activity; and endothelial-nitric oxide (NO) formation.

Recent study of DLBS2411 in healthy volunteers demonstrated the effective role and safety of DLBS2411 in suppressing intragastric acidity. Having such mechanisms of action, DLBS2411 is hypothesized to benefit in peptic ulcers.

DETAILED DESCRIPTION:
A total of 140 subjects will be allocated into 2 groups of treatment; each group will consist of 70 subjects with the treatment regimens:

Treatment I : 2 capsules of Omeprazole 20 mg, once daily and 1 placebo caplet of DLBS2411, twice daily Treatment II : 1 caplet of DLBS2411 250 mg, twice daily and 2 placebo capsules of omeprazole, once daily

DLBS2411 will be administered twice daily at least 30 minutes before morning and evening meals, while omeprazole, once daily before morning meals, for 8 weeks of study period.

The eligible subjects will receive either study medication (Treatment 1 or Treatment 2), for 8 weeks of treatment; and will be instructed to come to the clinic every 4-week interval throughout the study period.

Subjects will be evaluated for treatment efficacy at baseline and at interval of 4 weeks over the 8-week course of therapy.

The safety profile of study medication other than vital signs and adverse event will be measured at baseline and end of study. Vital signs and adverse event will be measured at baseline and every follow-up visit including end of study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-75 years old.
* Diagnosed as non-bleeding peptic ulcers who do not require endoscopic therapy, as confirmed by :

  * The presence of endoscopically confirmed gastric or duodenal ulcer(s) at size(s) of at least 3 mm or larger.
* Subjects with low-risk of recurrent bleeding, defined as both:

  * Complete Rockall score of ≤ 7.
  * Endoscopic stigmata (lesion) of grade II-C or III based on Forrest classification.
* Able to take oral medication.

Exclusion Criteria:

* For females of childbearing potential: pregnancy, breast-feeding, the intention of becoming pregnant during the study participation.

  * Patients must accept pregnancy tests during the trial if menstrual cycle is missed
  * Fertile patients must use a reliable and effective contraceptive
* History of or known or suspected Zollinger Ellison syndrome.
* History of endoscopic therapy for bleeding ulcer within the past 4 weeks.
* Indication for endoscopic hemostasis therapy.
* Presence of Helicobacter pylori infection
* History of or known coronary artery disease (CAD), congestive heart failure, pulmonary disease, and any other uncontrolled chronic diseases.
* History of or known gastrointestinal malignancy or ulcers associated to malignancy.
* Currently known being afflicted by serious infection(s).
* Inadequate liver function
* Inadequate renal function
* Subjects being under therapy with any herbal medicines.
* Known hypersensitivity or idiosyncratic reaction or adverse drug reactions to proton pump inhibitors (PPIs).
* Participation in any other clinical studies within 30 days prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-10; Primary Completion 2019-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Endoscopic ulcer healing rate | 8 weeks
  Endoscopic ulcer healing rate after 8 weeks of treatment. Ulcer healing rate is defined as the proportion of subjects with complete ulcer-healing (referring to S1 or S2 Scarring stage according to Sakita-Fukutomi classification) as confirmed by endoscopic finding.

SECONDARY OUTCOMES:
The improvement rate of each of gastric symptoms | 4 and 8 weeks
  The improvement rate of each of gastric symptoms at each of the follow-up visits (after 4 and 8 weeks of treatment):
  * abdominal or epigastric pain (middle or upper stomach)
  * nausea or vomiting,
  * bloating
The quality of ulcer healing | 8 weeks
  The quality of ulcer healing as measured by the levels of gastric mucosal bFGF (basic fibroblast growth factor) and COX-2 (cyclo-oxygenase), at baseline and Week 8 of treatment.
Mucosal thickness | 8 weeks
  Gastric mucosal thickness will be measured quantitatively as the expression of MUC5AC by immunohistochemistry (IHC) method, at baseline and Week 8 of treatment.
Patients' global evaluation for their symptoms | 4 and 8 weeks
  Patients' global evaluation for their symptoms categorized as: no improvement or slightly improved or moderately improved or markedly improved, at Week 4 and 8 (end of study).
Liver function | 8 weeks
  Liver function (serum ALT (alanine-aminotransferase), serum AST (aspartate-aminotransferase), alkaline phosphatase, total bilirubin) at baseline and at the end of study
Renal function | 8 weeks
  Renal function (serum creatinine and BUN (blood urea nitrogen) level) at baseline and at the end of study
Adverse events | 4 and 8 weeks
  Adverse event, will be observed throughout the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: IDN Wibawa Prof. DR. Dr., SpPD-KGEH, Principal Investigator — Division of Gastroenterohepatology Department of Internal Medicine Faculty of Medicine, University of Udayana Sanglah General Hospital
Locations (1):
- Division of Gastroenterohepatology Department of Internal Medicine Faculty of Medicine, University of Udayana Sanglah General Hospital, Denpasar, Bali, Indonesia